CLINICAL TRIAL: NCT01295164
Title: Feasibility of Measurement of High Order Aberrations in Late Stages Keratoconus by Using an Adaptive Optics Visual Simulator AOVIS-I
Brief Title: Measurement of High Order Aberrations in Late Stages Keratoconus
Acronym: VOPTICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10 214 03
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Keratoconus
Keywords: keratoconus, wave-front sensing technology, aberrometer
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): Measurement of aberrations in patients with keratoconus of grade 1
  Interventions: Device: classic aberrometer and aberrometer AOVIS-1
- Group 2 (Active Comparator): patients with keratoconus of grade 2
  Interventions: Device: classic aberrometer and aberrometer AOVIS-1
- Group 3 (Experimental): patients with keratoconus of grade 3
  Interventions: Device: Aberrometer AOVIS-I
- Group 4 (Experimental): patients with keratoconus of grade 4
  Interventions: Device: Aberrometer AOVIS-I

INTERVENTIONS:
Device: classic aberrometer and aberrometer AOVIS-1 — Measurement of aberrations in early stages (1 and 2) of keratoconus as compared aberrometer AOVIS-1 with a "classic aberrometer".
  Arms: Group 1; Group 2
Device: Aberrometer AOVIS-I — Measurement of aberrations in high stages (3 and 4) of keratoconus. Objective characterization of the optical quality of the patient eye by application of wave-front sensing technology in late stage keratoconus The complete procedure in one patient takes less than 5 minutes in only one consultation and is completely non invasive. The optical measurements only involve the use of low power infrared laser
  Arms: Group 3; Group 4

SUMMARY:
The instrument that will be used in the study is the Murcia monocular Adaptive Optics Visual simulator (AOVIS-I). The system provides an objective characterization of the optical quality of the patient's eye by application of wave-front sensing technology. The optical condition of every eye is represented by its wave aberration. This characterization overcomes the current description based only in refractive errors. This provides an accurate description of the optics of the eye based on the assessment of the whole set of ocular aberrations. The particular wave-front sensor is of a Hartmann-Shack type. One characteristics of this wave-front sensor is its high dynamic range allowing measuring highly aberrated eyes, such as patients with keratoconus.

DETAILED DESCRIPTION:
The complete procedure in one patient takes less than 5 minutes and is completely non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* to be able to understand an information and give a consent
* patients over 18
* patients with keratoconus
* affiliated to medical insurance.

Exclusion Criteria:

* non keratoconus patients
* patients under 18
* pregnant women or nursing mothers
* ocular surgery 90 days before inclusion
* ocular infection
* keratitis
* restless patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is to evaluate the AOVIS-I and its wave-front sensor with high dynamic range for measuring high-order aberrations in patients with late stages (3 and 4) of keratoconus | at the 1st day

SECONDARY OUTCOMES:
To evaluate the reliability of the measures in early stages (1 and 2) of keratoconus as compared with a "classic aberrometer". | at the 1st day
To describe the measures obtained in advanced stages (3 and 4) of keratoconus. | at the 1st day

CONTACTS AND LOCATIONS:
Overall Officials: Francois Malecaze, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hopstial Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No